CLINICAL TRIAL: NCT04881786
Title: The Effect of Orthodontic Forces on Calcitonin Gene-related Peptide Expression in Human Periodontal Ligament
Brief Title: Calcitonin Gene-related Peptide Expression in Human Periodontal Ligament
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institucion Universitaria Colegios de Colombia (Other)
Collaborators: Universidad Santo Tomas (Other)
Responsible Party: Principal Investigator, Javier Caviedes-Bucheli, Principal Investigator, Institucion Universitaria Colegios de Colombia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: JCB003
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: CGRP Expression in Human Periodontal Ligament
Keywords: Orthodontics forces; Calcitonin gene-related peptide; Periodontal ligament

STUDY DESIGN:
Intervention Model Description: from 90 premolars that were randomly divided into 3 groups of 30 premolars each, as follows: I) Untreated teeth control group (without orthodontic forces); II) Moderate force group; III) Severe force group. Teeth in moderate and severe orthodontic force groups were submitted to tipping and extrusion orthodontic movements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Untreated teeth control group (No Intervention): Premolars without orthodontic forces
- Moderate force group (Experimental): Premolars were submitted to tipping and extrusion orthodontic movements, the activation angle was 45º with a force of 56 g. Forces were measured with an orthodontic dynamometer. For 7 days
  Interventions: Device: Orthodontic forces
- Severe force group (Experimental): Premolars were submitted to tipping and extrusion orthodontic movements, the activation angle was 90º with a force of 224 g. Forces were measured with an orthodontic dynamometer. For 24 hours
  Interventions: Device: Orthodontic forces

INTERVENTIONS:
Device: Orthodontic forces — 56g force and 224g force
  Arms: Moderate force group; Severe force group

SUMMARY:
The purpose of this study was to quantify the effect of moderate and severe orthodontic forces on Calcitonin gene-related peptide expression in the healthy human periodontal ligament.

Methodology: 90 human periodontal ligament samples were obtained from healthy premolars where extraction was indicated for orthodontic reasons. Prior to extraction, teeth were divided into 3 groups of 30 samples each: I) Untreated teeth control group; II) Moderate force group: A 56 g force was applied to the premolars for 7 days; and III) Severe force group: A 224 g force was applied to the premolars for 24 hours. All periodontal ligament samples were processed and CGRP was measured by radioimmunoassay.

DETAILED DESCRIPTION:
An experimental study was performed according to Colombian Ministry of Health recommendations regarding ethical issues in research involving human tissue. Written informed consent was obtained from each of the patients participating in the study (18-27 years old, healthy, not medicated, and nonsmoking human donors, with premolars extraction indicated for orthodontic reasons). All teeth used were caries- and restoration-free with complete root development determined radiographically (and confirmed visually after extraction), without signs of periodontal disease or traumatic occlusion, and without previous orthodontic forces.

Experimental procedure Periodontal ligament samples were obtained from 90 premolars that were randomly divided into 3 groups of 30 premolars each, as follows: I) Untreated teeth control group (without orthodontic forces); II) Moderate force group; III) Severe force group. Teeth in moderate and severe orthodontic force groups were submitted to tipping and extrusion orthodontic movements.

Orthodontic forces were applied following the exact same methodology that was used in a previous study (15), in which, prior to orthodontic force application, the occlusal surface of the first mandibular molar was raised with a block of resin (Filtek Z350, 3M Espe, Seefeld, Germany) until the premolars were out of occlusion. A convertible standard buccal tube (Orthorganizer, Carlsbad, CA) was bonded over the buccal face of the first molar with resin (Light Bond, Reliance Orthodontic Products Inc, Itasca, IL). An MBT slot size 0.022 bracket (Ref. 702-393 MC, Orthorganizer) was bonded over the buccal face of the premolars. One 0.0017 x 0.025 in titanium molybdenum alloy (TMA) wire cantilever was inserted into each first molar tube and the wire was bent buccally to form a helix.

The cantilever was clinched to the distal end of the tube and exerted a tipping and extrusive force on the premolar. For the teeth in the moderate force group, the activation angle was 45º with a force of 56 g. For the severe force group, the activation angle was 90º with a force of 224 g. For both groups, forces were measured with an orthodontic dynamometer. Once the force was measured, the free-end of the sectional arch was hooked to the bracket with a metallic ligature. Seven days after, the ligature, the sectional arch, the tube, and the resin block were removed in order to perform the extraction procedure.

All teeth were anesthetized with 1.8 mL 4% prilocaine without vasoconstrictor by infiltrative injection for upper premolars and inferior alveolar nerve block injection for lower premolars. Adequate pulpal anesthesia was ascertained with a negative response to an electronic pulp vitality test.

Sample collection Teeth in the control and orthodontic forces group were extracted 10 min after anesthetic application with conventional methods and without excessive injury to the periodontal ligament. Immediately after extraction, PDL samples were obtained from the entire length of the root with a periodontal curette, placed on an Eppendorf tube, snap-frozen in liquid nitrogen, and kept at -70°C until use.

Radioimmunoassay (RIA) PDL samples were defrosted without thermal shock, dried on a filter, and individually weighed on an analytical balance. Neuropeptide was extracted by adding 150 µL of 0.5 mol L-1 acetic acid and double boiling in a thermostat bath for 30 min in accordance with previously reported protocols (9,12,15,18-21).

CGRP expression was determined by competition binding assays using a human CGRP-RIA kit from Phoenix Peptide Pharmaceutical (Ref. RK-015-02, Belmont, CA). Fifty µL of each sample solution were incubated in polypropylene tubes at room temperature for 20 h with 100 µL of primary antibody and 100 µL of different CGRP concentrations (10 pg mL-1 -1280 pg mL-1). Then, 50 µL of 125I-CGRP was added and left incubate for another 24 h. Bound fractions were precipitated by the addition of 100 µL of a secondary antibody (Goat Anti- Rabbit IgG serum), 100 µL of normal rabbit serum, and 500 µL of RIA buffer containing 1% polyethylene glycol 4000. After 2 h of incubation at room temperature, tubes were spun at 3000 rpm for 45 min at 4º C. The supernatants were decanted, and pellet radioactivity was read on a Gamma Counter (Gamma Assay LS 5500; Beckman, Fullerton, CA). Standard curves of authentic peptide were made in buffers identical to the tissue extracts on semi-log graph paper.

Finally, analysis of the binding data assessed the amount of CGRP present in every sample, using the percentage of maximum binding (B/B0%) calculated for each unknown sample, reading across the graph to the point of intersection with the calibration curve, where the corresponding X-axis coordinate is equivalent to the concentration of peptide in the assayed sample.

Statistical analysis Values are presented as CGRP concentration in pmol per mg of PDL. Mean, standard deviation, medians, and maximum/minimum values are presented for each group. Kruskal Wallis test was performed to establish statistically significant differences between groups (P<0.05). LSD posthoc comparisons were also performed.

ELIGIBILITY:
Inclusion Criteria:

- Premolars extraction indicated for orthodontic reasons with complete root development determined radiographically (and confirmed visually after extraction)

Exclusion Criteria:

* Medicated patients,
* Smokers patients,
* Premolars with caries or restorations,
* Premolars with signs of periodontal disease or traumatic occlusion,
* Premolars with previous orthodontic forces

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Calcitonin gene-related peptide in periodontal ligament | 24 hours stimulation and 7 days stimulation
  CGRP expression change in periodontal ligament

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Santo Tomas, Bucaramanga, Metropolitana, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beertsen W, McCulloch CA, Sodek J. The periodontal ligament: a unique, multifunctional connective tissue. Periodontol 2000. 1997 Feb;13:20-40. doi: 10.1111/j.1600-0757.1997.tb00094.x. No abstract available. PMID 9567922
- [Background] McCulloch CA, Lekic P, McKee MD. Role of physical forces in regulating the form and function of the periodontal ligament. Periodontol 2000. 2000 Oct;24:56-72. doi: 10.1034/j.1600-0757.2000.2240104.x. No abstract available. PMID 11276873
- [Background] Lekic P, McCulloch CA. Periodontal ligament cell population: the central role of fibroblasts in creating a unique tissue. Anat Rec. 1996 Jun;245(2):327-41. doi: 10.1002/(SICI)1097-0185(199606)245:23.0.CO;2-R. PMID 8769671
- [Background] Roberts WE, Goodwin WC Jr, Heiner SR. Cellular response to orthodontic force. Dent Clin North Am. 1981 Jan;25(1):3-17. PMID 6937399
- [Background] Sandy JR, Farndale RW, Meikle MC. Recent advances in understanding mechanically induced bone remodeling and their relevance to orthodontic theory and practice. Am J Orthod Dentofacial Orthop. 1993 Mar;103(3):212-22. doi: 10.1016/0889-5406(93)70002-6. PMID 8456777
- [Background] Caviedes-Bucheli J, Munoz HR, Azuero-Holguin MM, Ulate E. Neuropeptides in dental pulp: the silent protagonists. J Endod. 2008 Jul;34(7):773-88. doi: 10.1016/j.joen.2008.03.010. PMID 18570980
- [Background] Price TJ, Flores CM, Cervero F, Hargreaves KM. The RNA binding and transport proteins staufen and fragile X mental retardation protein are expressed by rat primary afferent neurons and localize to peripheral and central axons. Neuroscience. 2006 Sep 15;141(4):2107-16. doi: 10.1016/j.neuroscience.2006.05.047. Epub 2006 Jun 30. PMID 16809002
- [Background] Vandevska-Radunovic V. Neural modulation of inflammatory reactions in dental tissues incident to orthodontic tooth movement. A review of the literature. Eur J Orthod. 1999 Jun;21(3):231-47. doi: 10.1093/ejo/21.3.231. PMID 10407533
- [Background] Caviedes-Bucheli J, Azuero-Holguin MM, Correa-Ortiz JA, Aguilar-Mora MV, Pedroza-Flores JD, Ulate E, Lombana N, Munoz HR. Effect of experimentally induced occlusal trauma on substance p expression in human dental pulp and periodontal ligament. J Endod. 2011 May;37(5):627-30. doi: 10.1016/j.joen.2011.02.013. PMID 21496661
- [Background] Krishnan V, Davidovitch Z. On a path to unfolding the biological mechanisms of orthodontic tooth movement. J Dent Res. 2009 Jul;88(7):597-608. doi: 10.1177/0022034509338914. PMID 19641146
- [Background] Caviedes-Bucheli J, Azuero-Holguin MM, Gutierrez-Sanchez L, Higuerey-Bermudez F, Pereira-Nava V, Lombana N, Munoz HR. The effect of three different rotary instrumentation systems on substance P and calcitonin gene-related peptide expression in human periodontal ligament. J Endod. 2010 Dec;36(12):1938-42. doi: 10.1016/j.joen.2010.08.043. Epub 2010 Oct 15. PMID 21092809
- [Background] Caviedes-Bucheli J, Moreno JO, Ardila-Pinto J, Del Toro-Carreno HR, Saltarin-Quintero H, Sierra-Tapias CL, Macias-Gomez F, Ulate E, Lombana-Sanchez N, Munoz HR. The effect of orthodontic forces on calcitonin gene-related peptide expression in human dental pulp. J Endod. 2011 Jul;37(7):934-7. doi: 10.1016/j.joen.2011.03.035. Epub 2011 May 18. PMID 21689547